CLINICAL TRIAL: NCT02178839
Title: The Effect of Oral β- Glucan Supplement on Anthropometric Measurements, Appetite, Insulin Resistance, Liver Echogenicity and Enzymes in Non Alcoholic Fatty Liver Disease Treating With Hypocaloric Diet and Vitamin E
Brief Title: The Effect of Oral β- Glucan Supplement on Appetite and Insulin Resistance in Non Alcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: umsu.rec.1393.48
Record Dates: First submitted 2014-06-18; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Non Alcoholic Fatty Liver Disease(NAFLD); β- glucan; Appetite; Insulin Resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- β- glucan (Experimental): 8.5 g/d of Oat Supplement Containing 3g β- glucan
  Interventions: Dietary Supplement: β- glucan
- Maltodextrin (Placebo Comparator): 8.5 g/d Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: β- glucan — 8.5 g/d of Oat Supplement Containing 3g β- glucan
  Arms: β- glucan
Dietary Supplement: Maltodextrin — 8.5 g/d Maltodextrin
  Arms: Maltodextrin

SUMMARY:
The Objective of This Study is Evaluating the Effect of oral β- glucan Supplement on Anthropometric Measurements, Appetite, Insulin Resistance, Liver echogenicity and Enzymes in Non Alcoholic Fatty Liver Patients Treating with Hypocaloric Diet and Vitamin E.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non Alcoholic Fatty Liver Disease From Both Sex
* Age 18-55 years
* BMI more than 25 Kg/m2

Exclusion Criteria:

* Alcohol Consumption
* Pregnancy or lactation or menopause
* Being a professional athlete
* A history of cancer
* Risk of high blood pressure (in the case of drug use)
* Heart disease - cardiovascular, pulmonary, renal and diabetes
* Liver transplantation and other chronic or acute Liver diseases such as hepatitis B, C and liver infections
* The History of inherited disorders affecting the liver
* A history of autoimmune disease
* History of food allergies
* Taking certain medications such as blood pressure control, statins, insulin sensitivity enhancers and hepatotoxic drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Liver Echogenicity | 8 weeks
  Liver Echogenicity Describes by Grade,
Liver Enzymes | 8 weeks
  Enzymes ALP (Alkanin Phosphatase), ALT (Alanin Amino Transferase) and AST (Aspartat Amino Transferase)

SECONDARY OUTCOMES:
Anthropometric Measurement WHtR | 4 weeks, 8 weeks
  WHtR (waist to Height ratio)
Appetite | 4 weeks, 8 weeks
  NAS (numeric Analuge Scale) cm
Insulin Resistance | 8 weeeks
  Describe by HOMA-IR (Homeostasis Model Assessment of Insulin Resistance)
Anthropometric Measurement WC | 4weeks, 8 weeks
  WC (waist circumference) measures by "cm"
Anthropometric Measurement WHR | 4 weeks, 8 weeks
  WHR (waist to hip ratio)
Anthropometric Measurement BMI | 4 weeks, 8 weeks
  BMI (Body Mass Index) kg/m2
Peptide YY (PYY) Hormone | 8 weeks
  Elayza kit
Cholecystokinin (CKK) Hormone | 8 weeks
  Elayza kit
Fasting Blood Sugar | 8 weeks
  FBS (Fasting Blood Sugar) mmol/lit

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Alizadeh, PhD, Principal Investigator — Department of Nutrition, School of Medicine, Urmia University of Medical Sciences
Locations (1):
- Shekh-al- rais Clinic, Tabriz, Iran